CLINICAL TRIAL: NCT01923961
Title: Impact of an Increased Sodium Chloride Concentration in the Infusion Fluid of Predilution Hemodiafiltration on the Removal of Protein-Bound Uremic Toxins
Brief Title: Sodium Chloride and Protein-Bound Toxin Removal in Hemodiafiltration
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: EXcorLab GmbH (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: KSSA0113
Record Dates: First submitted 2013-08-10; First posted 2013-08-16 (Estimated); Results first posted 2019-01-16 (Actual); Last update posted 2019-01-16 (Actual); Status verified 2018-07

CONDITIONS: End-stage Renal Disease
Keywords: Maintenance hemodialysis or hemodiafiltration; >18 years; Stable condition
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — Renal Dialysis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- HDF NaCl, Then HD, Then Standard Pre-HDF (Experimental): Participants first receive hemodiafiltration with infusion of 5 M NaCl for 4 hours. After a washout period of 1 week, they then receive 4 hours of bicarbonate hemodialysis. After another washout period of 1 week, they reveive 4 hours of standard predilution hemodiafiltration.
  Interventions: Procedure: HDF NaCl; Procedure: Hemodialysis; Procedure: Standard Predilution Hemodiafiltration
- HD, Then Standard Pre-HDF, Then HDF NaCl (Experimental): Participants first receive bicarbonate hemodialysis for 4 hours. After a washout period of 1 week, they then receive 4 hours of standard predilution hemodiafiltration. After another washout period of 1 week, they reveive 4 hours of hemodiafiltration with infusion of 5 M NaCl.
  Interventions: Procedure: HDF NaCl; Procedure: Hemodialysis; Procedure: Standard Predilution Hemodiafiltration
- Standard Pre-HDF, Then HDF NaCl, Then HD (Experimental): Participants first receive standard predilution hemodiafiltration for 4 hours. After a washout period of 1 week, they then receive hemodiafiltration with infusion of 5 M NaCl 4 hours of. After another washout period of 1 week, they reveive 4 hours of bicarbonate hemodialysis.
  Interventions: Procedure: HDF NaCl; Procedure: Hemodialysis; Procedure: Standard Predilution Hemodiafiltration

INTERVENTIONS:
Procedure: HDF NaCl
  Other Names: Hemodialysis; Standard Predilution Hemodiafiltration
Procedure: Hemodialysis
  Other Names: Standard Predilution Hemodiafiltration; HDF NaCl
Procedure: Standard Predilution Hemodiafiltration
  Other Names: HDF NaCl; Hemodialysis

SUMMARY:
An increase of the free fraction may allow a better removal of of protein-bound uremic toxins during dialysis. During predilution hemodiafiltration, the sodium chloride (NaCl) concentration will be increased in the infusion fluid at a target NaCl concentration and the effect on the removal of protein-bound toxins will be determined. Comparisons will be made to standard hemodialysis and hemodiafiltration.

DETAILED DESCRIPTION:
Eight maintenance dialysis patients will be enrolled in a prospective, randomized, crossover trial. HD will be compared with online pre-dilution HDF and HDF at increased plasma ionic strength. The ionic strength will be increased using an infusion fluid with hypertonic [Na+] by isovolumetric adding of a 5000 mmol/L NaCl solution. Blood and dialysate flowrates (250 and 575 mL/min, respectively), treatment time (240 min), and high-flux dialyser (surface area 2.1 sqm, PUREMA H) will be always kept identical. Anticoagulation with standard or fractionated heparin will be unchanged adopted from the patients' routinely used regimen. In both HDF modes, the infusion flow rate will be 125 mL/min. In HDF at increased plasma ionic strength, the infusate [Na+] will be adjusted to approach 240 mmol/L in plasma entering the dialyser and the dialysate [Na+] will be set at the technically feasible minimum of 130 mmol/L. Blood samples will be drawn from the arterial and venous blood lines and, if applicable, from the blood tubing connecting the two dialyzers at 0, 15, 30, 60, 120, 180, and 240 min. Samples at 240 min will be drawn after reducing the blood flow rate to 50 mL/min for 30 s and the dialysate flow turned off. A fraction of the spent dialysate will be continuously collected.

Removal of the free and total fraction of para-cresyl sulfate and indoxyl sulfate will be determined by reduction ratios, dialytic clearances and mass in dialysate

Hemocompatibility will be assessed by WBC and platelet counts, free Hb, LDH, C5a and TAT. [Na+] will be monitored in both arterial (i.e. before NaCl infusion) and venous blood of the extracorporeal system.

ELIGIBILITY:
Inclusion Criteria:

* End-stage renal disease
* Maintenance hemodialysis or hemodiafiltration for more than 3 months
* Stable clinical condition
* > 18 years

Exclusion Criteria:

* Life expectancy less than 1 year
* Pregnancy
* Active infectious disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2013-08 (Actual); Primary Completion 2015-03-30 (Actual); Study Completion 2015-08-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Detlef H Krieter, MD, Principal Investigator — Wuerzburg University Hospital
Locations (1):
- Dialysis Center Elsenfeld, Elsenfeld, Bavaria, Germany

RESULTS

PARTICIPANT FLOW:
Groups:
- HDF NaCl Infusion, Then HD, Then Standard Pre-HDF: Participants first received hemodiafiltration with infusion of 5 M NaCl for 4 hours. After a washout period of 1 week, they then received 4 hours of bicarbonate hemodialysis. After another washout period of 1 week, they reveived 4 hours of standard predilution hemodiafiltration.
- HD, Then Standard Pre-HDF, Then HDF NaCl Infusion: Participants first received bicarbonate hemodialysis for 4 hours. After a washout period of 1 week, they then received 4 hours of standard predilution hemodiafiltration. After another washout period of 1 week, they reveived 4 hours of hemodiafiltration with infusion of 5 M NaCl.
- Standard Pre-HDF, Then HDF NaCl Infusion, Then HD: Participants first received standard predilution hemodiafiltration for 4 hours. After a washout period of 1 week, they then received 4 hours of hemodiafiltration with infusion of 5 M NaCl. After another washout period of 1 week, they reveived 4 hours of bicarbonate hemodialysis.
Period: First Intervention
Arm/Group | HDF NaCl Infusion, Then HD, Then Standard Pre-HDF | HD, Then Standard Pre-HDF, Then HDF NaCl Infusion | Standard Pre-HDF, Then HDF NaCl Infusion, Then HD
Started | 3 | 3 | 2
Completed | 3 | 3 | 2
Not Completed | 0 | 0 | 0
Period: Washout (1 Week)
Arm/Group | HDF NaCl Infusion, Then HD, Then Standard Pre-HDF | HD, Then Standard Pre-HDF, Then HDF NaCl Infusion | Standard Pre-HDF, Then HDF NaCl Infusion, Then HD
Started | 3 | 3 | 2
Completed | 3 | 3 | 2
Not Completed | 0 | 0 | 0
Period: Second Intervention
Arm/Group | HDF NaCl Infusion, Then HD, Then Standard Pre-HDF | HD, Then Standard Pre-HDF, Then HDF NaCl Infusion | Standard Pre-HDF, Then HDF NaCl Infusion, Then HD
Started | 3 | 3 | 2
Completed | 3 | 3 | 2
Not Completed | 0 | 0 | 0
Period: Washout (1 Week)
Arm/Group | HDF NaCl Infusion, Then HD, Then Standard Pre-HDF | HD, Then Standard Pre-HDF, Then HDF NaCl Infusion | Standard Pre-HDF, Then HDF NaCl Infusion, Then HD
Started | 3 | 3 | 2
Completed | 3 | 3 | 2
Not Completed | 0 | 0 | 0
Period: Third Intervention
Arm/Group | HDF NaCl Infusion, Then HD, Then Standard Pre-HDF | HD, Then Standard Pre-HDF, Then HDF NaCl Infusion | Standard Pre-HDF, Then HDF NaCl Infusion, Then HD
Started | 3 | 3 | 2
Completed | 3 | 3 | 2
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- HDF NaCl, Then HD, Then Standard Pre-HDF: Participants first received hemodiafiltration with infusion of 5 M NaCl for 4 hours. After a washout period of 1 week, they then received 4 hours of bicarbonate hemodialysis. After another washout period of 1 week, they reveived 4 hours of standard predilution hemodiafiltration.
- HD, Then Standard Pre-HDF, Then HDF NaCl: Participants first received bicarbonate hemodialysis for 4 hours. After a washout period of 1 week, they then received 4 hours of standard predilution hemodiafiltration. After another washout period of 1 week, they reveived 4 hours of hemodiafiltration with infusion of 5 M NaCl.
- Standard Pre-HDF, Then HDF NaCl, Then HD: Participants first received standard predilution hemodiafiltration for 4 hours. After a washout period of 1 week, they then received 4 hours of hemodiafiltration with infusion of 5 M NaCl. After another washout period of 1 week, they reveived 4 hours of bicarbonate hemodialysis.
- Total: Total of all reporting groups
Arm/Group | HDF NaCl, Then HD, Then Standard Pre-HDF | HD, Then Standard Pre-HDF, Then HDF NaCl | Standard Pre-HDF, Then HDF NaCl, Then HD | Total
Number analyzed (Participants) | 3 | 3 | 2 | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 2 | 2 | 1 | 5
  >=65 years | 1 | 1 | 1 | 3
Age, Continuous [Median (Full Range); unit: years] | 62 [46 to 78] | 62 [46 to 78] | 62 [46 to 78] | 62 [46 to 78]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 1 | 4
  Male | 1 | 2 | 1 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 3 | 3 | 2 | 8
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Germany | 3 | 3 | 2 | 8
Sodium Chloride (NaCl) Infusion [Count of Participants; unit: Participants] | 3 | 3 | 2 | 8

OUTCOME MEASURES:

1. Primary Outcome: Removal of Para-cresylsulfate
Description: Determination of reduction ratio, which is the ratio of a solute concentration in plasma at baseline and at the end of the intervention
Time Frame: 4 hours
Population: Per protocol population
Measure: Mean (Standard Deviation); unit: percentage of reduction
Groups:
- Hemodiafiltration, NaCl Infusion: 5 M NaCl solution will be infused to increase the NaCl concentration in the infusion fluid during predilution hemodiafiltration.
  5 M NaCl solution: Infusion of 5 M NaCl adjusted at target NaCl concentration in plasma.
- Hemodialysis: Standard bicarbonate high-flux hemodialysis
- Hemodiafiltration: Standard predilution Hemodiafiltration
Arm/Group | Hemodiafiltration, NaCl Infusion | Hemodialysis | Hemodiafiltration
Number analyzed (Participants) | 8 | 8 | 8
percentage of reduction | 42.0 (22.1) | 32.6 (18.5) | 33.6 (16.1)

2. Primary Outcome: Removal of Indoxylsulfate
Description: Determination of the reduction ratio, which is the ratio of a solute concentration in plasma at baseline and at the end of the intervention
Time Frame: 4 hours
Population: Per protocol analysis
Measure: Mean (Standard Deviation); unit: percentage of reduction
Arm/Group | Hemodiafiltration, NaCl Infusion | Hemodialysis | Hemodiafiltration
Number analyzed (Participants) | 8 | 8 | 8
percentage of reduction | 34.8 (23.5) | 26.5 (18.1) | 30.9 (23.9)

3. Secondary Outcome: Plasma Sodium Concentrations
Description: Maximum arterial sodium concentrations
Time Frame: 4 hours
Population: Per protocol analysis
Measure: Mean (Standard Deviation); unit: mval/l
Arm/Group | Hemodiafiltration, NaCl Infusion | Hemodialysis | Hemodiafiltration
Number analyzed (Participants) | 8 | 8 | 8
mval/l | 136 (3) | 133 (2) | 134 (2)

4. Secondary Outcome: Hemocompatibility
Description: Maximum free hemoglobin in plasma, which indicates hemolysis. Hemoglobin is released into plasma in case of red blood cell destruction.
Time Frame: 4 hours
Population: Per protocol analysis
Measure: Mean (Standard Deviation); unit: percentage of total hemoglobin
Arm/Group | Hemodiafiltration, NaCl Infusion | Hemodialysis | Hemodiafiltration
Number analyzed (Participants) | 8 | 8 | 8
percentage of total hemoglobin | 0.09 (0.04) | 0.07 (0.03) | 0.08 (0.02)

ADVERSE EVENTS:
Arm/Group | Hemodiafiltration, NaCl Infusion | Hemodialysis | Hemodiafiltration
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/8 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/8 | 0/8
Other Adverse Events (participants affected / at risk) | 0/8 | 0/8 | 0/8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No